CLINICAL TRIAL: NCT03359473
Title: A Randomized, Double-blind (Sponsor Unblind), Placebo-controlled, Multi-centred Phase IIa Study to Evaluate the Safety and Efficacy of 13 Weeks of Once Daily Oral Dosing of the Selective Androgen Receptor Modulator (SARM) GSK2881078 in Older Men and Post Menopausal Women With COPD and Muscle Weakness, Participating in Home Exercise
Brief Title: Study to Evaluate the Safety and Efficacy of 13 Weeks of the Selective Androgen Receptor Modulator (SARM) GSK2881078 in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200182; 2017-001148-37 (EudraCT Number)
Record Dates: First submitted 2017-11-22; First posted 2017-12-02 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-06

CONDITIONS: Cachexia
Keywords: GSK2881078; COPD; muscle weakness; post-menopausal; selective androgen receptor modulator
MeSH Terms: conditions — Cachexia; Pulmonary Disease, Chronic Obstructive; Muscle Weakness | interventions — GSK2881078

STUDY DESIGN:
Intervention Model Description: Study treatment will consist of two dosing cohorts: Cohort 1 will comprise of male subjects randomized to receive either placebo or 2 milligrams (mg) of GSK2881078 and Cohort 2 will comprise of post-menopausal female subjects randomized to receive either placebo or 1 mg of GSK2881078.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Male subjects receiving GSK2881078-Cohort 1 (Experimental): Male subjects between the age of 50 and 75 years will be administered GSK2881078 at a dose of 2 mg once daily by the oral route.
  Interventions: Drug: GSK2881078
- Male subjects receiving Placebo-Cohort 1 (Placebo Comparator): Male subjects between the age of 50 and 75 years will be administered GSK2881078 matching placebo once daily by the oral route.
  Interventions: Drug: Matching Placebo
- Female subjects receiving GSK2881078-Cohort 2 (Experimental): Post-menopausal female subjects between the age of 50 and 75 years will be administered GSK2881078 at a dose of 1 mg once daily by the oral route.
  Interventions: Drug: GSK2881078
- Female subjects receiving Placebo-Cohort 2 (Placebo Comparator): Post-menopausal female subjects between the age of 50 and 75 years will be administered GSK2881078 matching placebo once daily by the oral route.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: GSK2881078 — GSK2881078 will be available as capsules for oral administration. GSK2881078 will be administered once daily by the oral route at a dose of 1 mg and 2mg to post-menopausal female subjects and male subjects, respectively.
  Arms: Female subjects receiving GSK2881078-Cohort 2; Male subjects receiving GSK2881078-Cohort 1
Drug: Matching Placebo — Subjects will be administered two capsules of GSK2881078 matching placebo once daily by the oral route.
  Arms: Female subjects receiving Placebo-Cohort 2; Male subjects receiving Placebo-Cohort 1

SUMMARY:
Impaired physical function and muscle dysfunction are a major consequence of COPD, which may be associated with increased mortality, poor quality of life and increased health care use. This is a randomized, placebo-controlled, double-blind, parallel group study to evaluate the safety and tolerability of GSK2881078, an SARM over 13 weeks of dosing in older male subjects and post-menopausal female subjects with COPD and muscle weakness. This study will also assess the effect of GSK2881078 on physical strength and function after 13 weeks of treatment. Approximately 100 subjects with COPD and muscle weakness will be randomized into two cohorts of 50 male subjects and 50 female subjects. Within each cohort, subjects will be randomized to receive GSK2881078 or placebo in a ratio of 1:1. All subjects will participate in a standardized home exercise program, which will consist of daily walking, along with several resistance or weight-bearing exercises, such as bicep curls, upright rows, step ups and a sit-to-stand maneuver. The study will consist of a screening/Baseline period of up to 30 days, a 13-week treatment period and a post-treatment follow-up period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 50 to 75 years of age inclusive, at the time of signing the informed consent.
* Male and/or female subjects will be included. a) A male subject with a partner who is a woman of child bearing potential (WOCPB) must agree to use contraception during the treatment period and until at least 5 half-lives of study medication have passed after the last ingested dose [125 days, corresponding to time needed to eliminate study treatment for both genotoxic and teratogenic study treatments plus an additional 90 days (a spermatogenesis cycle) for study treatments with genotoxic potential] after the last dose of study treatment and refrain from donating sperm during this period. b) A female subject is eligible to participate if she is post-menopausal and not a WOCBP.
* Confirmed diagnosis of COPD in accordance with the American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria with a post-bronchodilator FEV1/forced vital capacity (FVC) <0.70 and 30% <= FEV1% predicted <=65% of predicted normal value calculated at Screen using the Quanjer reference equation.
* SPPB with ALL of the following: Timed chair stand score >=1 and <=3; No score of "0" on any component of the SPPB (that is, gait speed, balance, or timed chair stand).
* Body Mass Index (BMI) within the range 18-32 kilogram per meter square (kg/m^2) (inclusive), where BMI = (weight in kg)/(height in meters)^2
* Current smokers or former smokers with a cigarette smoking history of >=10 pack years (1 pack year =20 cigarettes smoked per day for 1 year or equivalent). Former smokers are defined as those who have stopped smoking for at least 6 months prior to Baseline.
* Subjects must be able to read and write in the language used for the provided electronic diary and be able to operate an electronic device to a level that allows them to complete an electronic diary on a daily basis.
* Subjects participating in a structured exercise program must be willing to convert their current exercise program to the home exercise program used in this study.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and protocol.

Exclusion Criteria:

* Subjects with a history of myocardial infarction, angina, congestive heart failure exacerbation, hospitalization for cardiac etiology, stroke or transient ischemic attack in the past 12 months.
* Neurologic, musculoskeletal, osteoarthritis, or any other condition that in the opinion of the investigator limits subject's ability to complete study physical assessments.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a history of cholecystectomy.
* Subjects with a history of malignancy that is not in complete remission for at least 2 years or 1 year for non-melanoma skin carcinoma.
* Subjects with a family history of early onset prostate cancer or familial prostate cancer (multiple family members).
* Diseases known to cause malabsorption of protein or energy, such as inflammatory bowel disease, celiac disease, pancreatic insufficiency, etc.
* Current or planned administration of cholestyramine or strong oral or injectable cytochrome P-450 isoenzyme 3A4 (CYP3A4) inducers.
* Current or planned use of any prescription drugs known to affect muscle mass, including androgen supplements, anti-androgens (such as luteinizing hormone-releasing hormone [LHRH] agonists), anti-estrogens (tamoxifen, etc.), recombinant growth hormone, megesterol, etc.
* Use of oral steroids concurrently or within 4 weeks preceding the screening visit.
* The subject has participated in a clinical trial and has received an investigational product within the following time-period prior to randomization in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Subjects with values outside the specified ranges for the following Key Clinical Laboratory Tests must be excluded from the study: a) Renal function: Glomerular Filtration Rate (GFR) <30 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2). Subjects receiving dialysis are excluded from this study. b) Metabolic-glycated hemoglobin (HbA1c) >7.5%. c) ALT >2 times upper limit of normal (ULN) and bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). d) Hematology - Hemoglobin <10.0 grams per deciliter (g/dL) at screening. e) Prostate Specific Antigen (PSA) >4.0 nanograms per milliliter (ng/mL).
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* QT interval corrected for heart rate by Bazett's formula (QTcB) or QT interval corrected for heart rate by Fridericia's formula (QTcF) >450 milliseconds (msec) or QT interval corrected for heart rate (QTc) >480 msec in subjects with Bundle Branch Block based on a single ECG.
* A positive test for human immunodeficiency virus (HIV) antibody.
* More than two moderate/severe COPD exacerbations within the past year. Exacerbation is defined as worsening of two or more of the following major symptoms: dyspnea, sputum volume, sputum purulence OR worsening of any one major symptom together with at least one of the following additional symptoms: sore throat, colds (nasal discharge and/or nasal congestion), fever >37.5 degree Celsius without any explained cause, increased cough, increased wheeze. A moderate exacerbation is defined as an exacerbation that requires treatment with antibiotics and/or oral steroids. A severe exacerbation is defined as an event that is additionally associated with hospitalization or emergency room visit.
* Any moderate/severe COPD exacerbation in the 4 weeks preceding the screening visit.
* Subjects on long-term oxygen therapy (LTOT), defined as prescribed continuous oxygen use for >14 hours/day.
* Clinically diagnosed history of drug or alcohol abuse within 5 years prior to randomization.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Participation in a formal pulmonary rehabilitation exercise program outside or inside the home, either currently or completed within the previous 6 months.
* For subjects who opt to have magnetic resonance imaging (MRI) at participating study sites, there must be no contraindications to MRI, for example known claustrophobia or a pacemaker. Specific MRI contraindications will be determined by the type of MRI scanner available at each site and study personnel should confirm local eligibility requirements.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (5):
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
- Germany (2):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
- United Kingdom (4):
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Harefield, Middlesex
  - GSK Investigational Site, London
  - GSK Investigational Site, London, Greater London

REFERENCES:
- [Derived] Tabberer M, Williamson N, Tatlock S, Gater A, Grimes R, Akinseye C, Neil D, Mahon-Smith A, Nelsen L. Qualitative interviews of patients with COPD and muscle weakness enrolled in a clinical trial evaluating a new anabolic treatment: patient perspectives of disease experience, trial participation and outcome assessments. J Patient Rep Outcomes. 2024 Apr 20;8(1):45. doi: 10.1186/s41687-024-00712-0. PMID 38641716
- [Derived] Mohan D, Rossiter H, Watz H, Fogarty C, Evans RA, Man W, Tabberer M, Beerahee M, Kumar S, Millns H, Thomas S, Tal-Singer R, Russell AJ, Holland MC, Akinseye C, Neil D, Polkey MI. Selective androgen receptor modulation for muscle weakness in chronic obstructive pulmonary disease: a randomised control trial. Thorax. 2023 Mar;78(3):258-266. doi: 10.1136/thorax-2021-218360. Epub 2022 Oct 25. PMID 36283827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase II, double-blind, randomized, multicenter study to evaluate the safety and efficacy of GSK2881078 over 13 weeks of once daily oral dosing, first time administered in older men and post-menopausal female participants with chronic obstructive pulmonary disease (COPD) and muscle weakness, participating in home exercise.
Pre-assignment Details: A total of 200 participants were screened and 97 participants were enrolled in this study. Of which, 96 participants were randomized and received the study treatment. The remaining 1 participant was randomized without fulfilling the inclusion and exclusion criteria and therefore did not receive study medication.
Groups:
- Placebo- Female Participants: Post-menopausal female participants, 50 to 75 years of age, were administered orally two capsules of GSK2881078 matching placebo once daily over 13 weeks.
- GSK2881078 1.0 mg- Female Participants: Post-menopausal female participants, 50 to 75 years of age, were administered orally two capsules of GSK2881078 of a unit dose strength 0.5 milligram (mg) once daily over 13 weeks.
- Placebo- Male Participants: Male participants, 50 to 75 years of age, were administered orally two capsules of GSK2881078 matching placebo once daily over 13 weeks.
- GSK2881078 2.0 mg- Male Participants: Male participants, 50 to 75 years of age, were administered orally two capsules of GSK2881078 of a unit dose strength 1.0 mg once daily over 13 weeks.
Period: Overall Study
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Started | 23 | 24 | 24 | 25
Completed | 21 | 18 | 18 | 20
Not Completed | 2 | 6 | 6 | 5
Not completed — Adverse Event | 0 | 2 | 5 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0
Not completed — Protocol-defined stopping criteria | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants | Total
Number analyzed (Participants) | 23 | 24 | 24 | 25 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (7.16) | 64.2 (7.93) | 64.0 (7.27) | 67.2 (6.08) | 65.1 (7.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 0 | 0 | 47
  Male | 0 | 0 | 24 | 25 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 2 | 2 | 5
  White-White/Caucasian/European Heritage | 23 | 23 | 22 | 23 | 91

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in a seated position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Safety Population comprised of all randomized participants who received at least one dose of study medication. This population was based on the treatment the participant received.
Time Frame: Baseline (Day 1, Pre-dose), Days 14, 28, 56 and 90
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 22 | 23 | 23 | 24
Millimeters of mercury
  SBP,Day 14,n=22,23,23,24 | 3.0 (19.63) | 2.1 (11.03) | -2.1 (9.33) | 3.1 (11.65)
  SBP,Day 28,n=22,20,23,24: number analyzed (Participants) | 22 | 20 | 23 | 24
  SBP,Day 28,n=22,20,23,24 | 3.7 (12.76) | -0.1 (12.82) | 2.6 (14.39) | 5.8 (9.49)
  SBP,Day 56,n=21,19,20,21: number analyzed (Participants) | 21 | 19 | 20 | 21
  SBP,Day 56,n=21,19,20,21 | 3.3 (14.96) | 7.8 (16.38) | -2.4 (17.68) | 1.3 (9.12)
  SBP,Day 90,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  SBP,Day 90,n=21,18,18,20 | 1.0 (14.23) | 7.6 (15.56) | -4.2 (18.52) | 5.8 (18.61)
  DBP,Day 14,n=22,23,23,24 | 1.9 (6.88) | 1.1 (6.93) | -3.4 (6.20) | -0.4 (7.47)
  DBP,Day 28,n=22,20,23,24: number analyzed (Participants) | 22 | 20 | 23 | 24
  DBP,Day 28,n=22,20,23,24 | 3.6 (7.08) | 1.4 (7.58) | 0.7 (7.90) | 1.0 (5.36)
  DBP,Day 56,n=21,19,20,21: number analyzed (Participants) | 21 | 19 | 20 | 21
  DBP,Day 56,n=21,19,20,21 | 2.1 (7.00) | 2.9 (6.07) | -2.5 (10.38) | -1.6 (8.16)
  DBP,Day 90,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  DBP,Day 90,n=21,18,18,20 | -1.0 (6.47) | 2.9 (8.37) | -0.1 (12.98) | 0.6 (6.95)

2. Primary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured in a seated position with a completely automated device. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 14, 28, 56 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 22 | 23 | 23 | 24
Beats per minute
  Day 14,n=22,23,23,24 | -0.7 (9.79) | 3.3 (9.16) | 1.7 (10.61) | -0.4 (6.60)
  Day 28,n=22,20,23,24: number analyzed (Participants) | 22 | 20 | 23 | 24
  Day 28,n=22,20,23,24 | 2.2 (8.11) | 2.1 (9.64) | 4.6 (10.71) | -1.7 (10.71)
  Day 56,n=21,19,20,21: number analyzed (Participants) | 21 | 19 | 20 | 21
  Day 56,n=21,19,20,21 | 0.2 (8.87) | -1.0 (8.81) | 2.8 (7.17) | 0.2 (6.36)
  Day 90,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90,n=21,18,18,20 | 1.1 (7.99) | 2.3 (10.34) | 7.4 (10.23) | -0.6 (8.17)

3. Primary Outcome: Change From Baseline in PR Interval, QRS Duration, QT Interval, QT Interval Corrected for Heart Rate by Fridericia's Formula (QTcF) and QT Interval Corrected for Heart Rate by Bazett's Formula (QTcB)
Description: Twelve-lead electrocardiograms (ECG) were obtained using an automated ECG machine to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 14, 28, 56 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 22 | 23 | 23 | 24
Milliseconds
  PR interval,Day 14,n=22,23,22,24: number analyzed (Participants) | 22 | 23 | 22 | 24
  PR interval,Day 14,n=22,23,22,24 | -1.303 (9.9261) | -0.377 (7.2588) | -2.455 (12.6556) | -2.875 (24.3370)
  PR interval,,Day 28,n=22,20,22,24: number analyzed (Participants) | 22 | 20 | 22 | 24
  PR interval,,Day 28,n=22,20,22,24 | -0.061 (7.9340) | -4.717 (19.3177) | -2.333 (17.5966) | 4.139 (15.5796)
  PR interval,,Day 56,n=21,19,20,21: number analyzed (Participants) | 21 | 19 | 20 | 21
  PR interval,,Day 56,n=21,19,20,21 | 1.302 (12.1220) | 0.596 (6.5250) | 0.483 (7.5436) | 10.444 (27.5133)
  PR interval,,Day 90,n=21,18,17,20: number analyzed (Participants) | 21 | 18 | 17 | 20
  PR interval,,Day 90,n=21,18,17,20 | -0.270 (9.3111) | -6.167 (28.9117) | -3.373 (9.6845) | 3.033 (20.7947)
  QRS Duration,Day 14,n=22,23,23,24 | 4.364 (22.8107) | 1.362 (10.4736) | -0.464 (7.4791) | 1.167 (4.1772)
  QRS Duration,Day 28,n=22,20,23,24: number analyzed (Participants) | 22 | 20 | 23 | 24
  QRS Duration,Day 28,n=22,20,23,24 | 1.000 (7.7014) | 6.200 (28.2707) | -1.478 (5.5047) | -0.542 (3.3547)
  QRS Duration,Day 56,n=21,19,20,21: number analyzed (Participants) | 21 | 19 | 20 | 21
  QRS Duration,Day 56,n=21,19,20,21 | -0.095 (5.9639) | 1.842 (5.4096) | -1.100 (4.9631) | -0.413 (4.6271)
  QRS Duration,Day 90,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  QRS Duration,Day 90,n=21,18,18,20 | -2.397 (14.1494) | -2.444 (4.5360) | 1.333 (25.4163) | 1.333 (6.3005)
  QT Interval,Day 14,n=22,23,23,24 | 0.576 (19.8239) | -14.290 (17.7216) | -0.638 (22.5431) | -0.597 (15.5697)
  QT Interval,Day 28,n=22,20,23,24: number analyzed (Participants) | 22 | 20 | 23 | 24
  QT Interval,Day 28,n=22,20,23,24 | -1.333 (23.5300) | -16.133 (26.2775) | -4.203 (23.3733) | -1.750 (22.6539)
  QT Interval,Day 56,n=21,19,20,21: number analyzed (Participants) | 21 | 19 | 20 | 21
  QT Interval,Day 56,n=21,19,20,21 | -0.127 (13.5567) | -13.947 (18.3657) | -1.533 (20.5897) | -1.857 (14.6881)
  QT Interval,Day 90,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  QT Interval,Day 90,n=21,18,18,20 | 4.063 (16.9160) | -16.352 (20.7511) | -4.574 (17.1825) | -5.167 (17.7759)
  QTcF Interval,Day 14,n=21,21,21,21: number analyzed (Participants) | 21 | 21 | 21 | 21
  QTcF Interval,Day 14,n=21,21,21,21 | 1.749 (11.7762) | -7.143 (9.2710) | -1.235 (11.3507) | -2.698 (9.7085)
  QTcF Interval,Day 28,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  QTcF Interval,Day 28,n=21,19,21,21 | 0.362 (15.7742) | -12.930 (11.7707) | -0.489 (10.5492) | -4.340 (12.8445)
  QTcF Interval,Day 56,n=20,18,18,18: number analyzed (Participants) | 20 | 18 | 18 | 18
  QTcF Interval,Day 56,n=20,18,18,18 | 1.333 (8.5039) | -12.222 (10.2975) | 1.093 (10.0462) | -3.357 (10.5127)
  QTcF Interval,Day 90,n=20,17,18,17: number analyzed (Participants) | 20 | 17 | 18 | 17
  QTcF Interval,Day 90,n=20,17,18,17 | 3.600 (10.3526) | -12.627 (11.5776) | 2.657 (12.2002) | -11.804 (11.7207)
  QTcB Interval,Day 14,n=4,5,4,7: number analyzed (Participants) | 4 | 5 | 4 | 7
  QTcB Interval,Day 14,n=4,5,4,7 | -4.333 (26.2100) | 2.193 (12.5624) | 12.917 (13.6582) | 0.571 (11.0180)
  QTcB Interval,Day 28,n=4,3,4,7: number analyzed (Participants) | 4 | 3 | 4 | 7
  QTcB Interval,Day 28,n=4,3,4,7 | -1.167 (12.1549) | 13.667 (24.7678) | -7.667 (8.8192) | -10.238 (11.6678)
  QTcB Interval,Day 56,n=3,3,4,6: number analyzed (Participants) | 3 | 3 | 4 | 6
  QTcB Interval,Day 56,n=3,3,4,6 | -13.556 (11.3741) | -7.667 (9.7125) | 13.417 (8.0017) | -9.500 (7.2411)
  QTcB Interval,Day 90,n=3,3,2,6: number analyzed (Participants) | 3 | 3 | 2 | 6
  QTcB Interval,Day 90,n=3,3,2,6 | 1.333 (15.9199) | -13.111 (3.0972) | 32.000 (1.4142) | -10.278 (9.6088)

4. Primary Outcome: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Hematology Parameters
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin (Hb), lymphocyte count (Lympho), neutrophil count (Neutro) and platelet count (PC). The laboratory parameters were graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Only those participants with increase to grade 3 and increase to grade 4 are presented.
Time Frame: Baseline (Day 1, Pre-dose) and up to Day 132
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 23 | 22 | 24 | 25
Participants
  Hb, Anemia, increase to Grade 3 | 0 | 0 | 0 | 0
  Hb, Anemia, increase to Grade 4 | 0 | 0 | 0 | 0
  Hb, Hb increased, increase to Grade 3 | 0 | 0 | 0 | 0
  Hb, Hb increased, increase to Grade 4 | 0 | 0 | 0 | 0
  Lympho, Lymph count decreased, increase to Grade 3 | 0 | 0 | 0 | 0
  Lympho, Lymph count decreased, increase to Grade 4 | 0 | 0 | 0 | 0
  Lympho, Lymph count increased, increase to Grade 3 | 0 | 0 | 0 | 0
  Lympho, Lymph count increased, increase to Grade 4 | 0 | 0 | 0 | 0
  Neutro,Neutro count decreased,increase to Grade 3 | 0 | 0 | 0 | 0
  Neutro,Neutro count decreased,increase to Grade 4 | 0 | 0 | 0 | 0
  PC, PC decreased,increase to Grade 3 | 0 | 0 | 0 | 0
  PC, PC decreased,increase to Grade 4 | 0 | 0 | 0 | 0
  PC, PC increased,increase to Grade 3 | 0 | 0 | 0 | 0
  PC, PC increased,increase to Grade 4 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Grade Increase Post-Baseline Relative to Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST), bilirubin (Bil),calcium (Ca), cholesterol (Chol), creatinine (Creat), glucose(Gl), phosphate (Phos), potassium (Pot) and sodium (Sod). The laboratory parameters were graded according to NCI-CTCAE version 4.03. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Values (Hyper and hypo) for Ca, Gl, Pot, Phos and Sod is presented. Only those participants with increase to grade 3 and increase to grade 4 are presented.
Time Frame: Baseline (Day 1, Pre-dose) and up to Day 132
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 23 | 22 | 24 | 25
Participants
  ALT, ALT increased, increase to Grade 3 | 0 | 1 | 0 | 1
  ALT, ALT increased, increase to Grade 4 | 0 | 0 | 0 | 0
  ALP, ALP increased, increase to Grade 3 | 0 | 0 | 0 | 0
  ALP, ALP increased, increase to Grade 4 | 0 | 0 | 0 | 0
  AST, AST increased, increase to Grade 3 | 0 | 0 | 0 | 0
  AST, AST increased, increase to Grade 4 | 0 | 0 | 0 | 0
  Bil, Blood Bil increased, increase to Grade 3 | 0 | 0 | 0 | 0
  Bil, Blood Bil increased, increase to Grade 4 | 0 | 0 | 0 | 0
  Ca, Hyper,increase to Grade 3 | 0 | 0 | 0 | 0
  Ca, Hyper,increase to Grade 4 | 0 | 0 | 0 | 0
  Ca, Hypo,increase to Grade 3 | 0 | 0 | 0 | 0
  Ca, Hypo,increase to Grade 4 | 0 | 0 | 0 | 0
  Chol, Chol high,increase to Grade 3 | 0 | 0 | 0 | 0
  Chol, Chol high,increase to Grade 4 | 0 | 0 | 0 | 0
  Creat, Creat increased,increase to Grade 3 | 0 | 0 | 0 | 0
  Creat, Creat increased,increase to Grade 4 | 0 | 0 | 0 | 0
  Gl, Hyper,increase to Grade 3 | 0 | 0 | 0 | 1
  Gl, Hyper,increase to Grade 4 | 0 | 0 | 0 | 0
  Gl, Hypo,increase to Grade 3 | 0 | 0 | 0 | 0
  Gl, Hypo,increase to Grade 4 | 0 | 0 | 0 | 0
  Phos, Hyper,increase to Grade 3 | 0 | 0 | 0 | 0
  Phos, Hyper,increase to Grade 4 | 0 | 0 | 0 | 0
  Phos, Hypo,increase to Grade 3 | 0 | 0 | 0 | 0
  Phos, Hypo,increase to Grade 4 | 0 | 0 | 0 | 0
  Pot, Hyper,increase to Grade 3 | 0 | 0 | 0 | 0
  Pot, Hyper,increase to Grade 4 | 0 | 0 | 0 | 0
  Pot, Hypo,increase to Grade 3 | 0 | 0 | 1 | 0
  Pot, Hypo,increase to Grade 4 | 0 | 0 | 0 | 0
  Sod, Hyper,increase to Grade 3 | 0 | 0 | 0 | 0
  Sod, Hyper,increase to Grade 4 | 0 | 0 | 0 | 0
  Sod, Hypo,increase to Grade 3 | 2 | 0 | 0 | 0
  Sod, Hypo,increase to Grade 4 | 0 | 0 | 0 | 0

6. Primary Outcome: Change From Baseline in Urinalysis Parameter; Specific Gravity: Placebo-Female Participants
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine, indicated as ratio of urine density to water density. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 28, 56 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo- Female Participants
Number analyzed (Participants) | 21
Ratio
  Day 28,n=1: number analyzed (Participants) | 1
  Day 28,n=1 | 0.0030 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 56,n=1: number analyzed (Participants) | 1
  Day 56,n=1 | 0.0020 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 90,n=21 | -0.0006 (0.00612)

7. Primary Outcome: Change From Baseline in Urinalysis Parameter; Specific Gravity: GSK2881078 1.0 mg- Female Participants
Description: as for outcome 6
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GSK2881078 1.0 mg- Female Participants
Number analyzed (Participants) | 18
Ratio
  Day 14,n=1: number analyzed (Participants) | 1
  Day 14,n=1 | 0.000 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 90,n=18 | 0.0049 (0.00711)

8. Primary Outcome: Change From Baseline in Urinalysis Parameter; Specific Gravity: Male Participants
Description: as for outcome 6
Time Frame: Baseline (Day 1, Pre-dose), Days 28 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 19 | 20
Ratio
  Day 28,n=1,1: number analyzed (Participants) | 1 | 1
  Day 28,n=1,1 | -0.0080 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 0.0040 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 90,n=19,20 | 0.0017 (0.00870) | 0.0018 (0.00610)

9. Primary Outcome: Change From Baseline in Urinalysis Parameter; Potential of Hydrogen (pH): Placebo- Female Participants
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 28, 56 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo- Female Participants
Number analyzed (Participants) | 21
pH
  Day 28,n=1: number analyzed (Participants) | 1
  Day 28,n=1 | 0.0000 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 56,n=1: number analyzed (Participants) | 1
  Day 56,n=1 | -0.5000 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 90,n=21 | 0.0000 (0.80623)

10. Primary Outcome: Change From Baseline in Urinalysis Parameter; pH: GSK2881078 1.0 mg- Female Participants
Description: as for outcome 9
Time Frame: Baseline (Day 1, Pre-dose), Days 14 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | GSK2881078 1.0 mg- Female Participants
Number analyzed (Participants) | 18
pH
  Day 14,n=1: number analyzed (Participants) | 1
  Day 14,n=1 | 1.0000 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 90,n=18 | -0.1111 (0.60768)

11. Primary Outcome: Change From Baseline in Urinalysis Parameter; pH: Male Participants
Description: as for outcome 9
Time Frame: Baseline (Day 1, Pre-dose), Days 28 and 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 19 | 20
pH
  Day 28,n=1,1: number analyzed (Participants) | 1 | 1
  Day 28,n=1,1 | 1.0000 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 0.5000 (NA) — Standard deviation could not be calculated as a single participant was analyzed.
  Day 90,n=19,20 | -0.1579 (0.72749) | 0.3000 (0.71451)

12. Primary Outcome: Number of Participants With Urinalysis Dipstick Results Post-Baseline Relative to Baseline
Description: Urine samples were collected to analyze parameters including glucose, occult blood (OB) and protein levels by dipstick. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as increase to trace, increase to 1+ (low concentrations present), increase to 2+ (moderate concentrations present) and increase to 3+ (high concentrations present) indicating proportional concentrations in the urine sample. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data for worst-case post-Baseline relative to Baseline is presented.
Time Frame: Baseline (Day 1, Pre-dose) and up to Day 132
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 23 | 21 | 23 | 24
Participants
  Glucose: increase to trace | 0 | 0 | 1 | 0
  Glucose: increase to 1+ | 0 | 0 | 0 | 0
  Glucose: increase to 2+ | 0 | 0 | 0 | 0
  Glucose: increase to 3+ | 0 | 0 | 0 | 1
  OB: increase to trace | 1 | 0 | 1 | 1
  OB: increase to 1+ | 1 | 1 | 1 | 0
  OB: increase to 2+ | 1 | 2 | 0 | 0
  OB: increase to 3+ | 0 | 0 | 0 | 1
  Protein: increase to trace | 2 | 2 | 3 | 6
  Protein: increase to 1+ | 0 | 3 | 1 | 3
  Protein: increase to 2+ | 0 | 1 | 0 | 1
  Protein: increase to 3+ | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. Number of participants who had SAEs and non-SAEs are presented.
Time Frame: Up to Day 132
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 23 | 24 | 24 | 25
Participants
  Non-SAEs | 15 | 18 | 13 | 17
  SAEs | 1 | 2 | 2 | 0

14. Primary Outcome: Percentage Change From Baseline in Maximum Leg Press Strength Following 1 Repetition Maximum (1-RM) at Day 28
Description: Lower extremity strength was measured as 1-RM on a leg press device. Participants continued with a one set of 5 to 10 repetitions of lifting weights using 40 to 60% of estimated maximum, after warm up. Participants, then lifted progressively heavier weights in steps, with each step separated by an appropriate rest period, until participant could not complete the lift. The last successfully completed lift was recorded as the 1-RM. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Percentage change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value]. Adjusted means and standard error (SE) are presented. Analysis Population comprised of the participants in the 'All Participants (all randomized participants who received at least one dose of study medication)' Population having Baseline and at least one post-Baseline assessment of the treatment the participant was randomized to.
Time Frame: Baseline (Day 1, Pre-dose), Day 28
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 20 | 22 | 23
Percentage change | 4.82 (2.406) | 9.34 (2.459) | 1.55 (2.940) | 9.35 (2.848)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 4.53, 90% CI 2-sided [-1.30 to 10.36] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and Baseline leg press strength, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 7.80, 90% CI 2-sided [0.83 to 14.76] — [estimate comment as in outcome 14, analysis 1]

15. Primary Outcome: Percentage Change From Baseline in Maximum Leg Press Strength Following 1 Repetition Maximum (1-RM) at Day 56
Description: Lower extremity strength was measured as 1-RM on a leg press device. Participants continued with a one set of 5 to 10 repetitions of lifting weights using 40 to 60% of estimated maximum, after warm up. Participants, then lifted progressively heavier weights in steps, with each step separated by an appropriate rest period, until participant could not complete the lift. The last successfully completed lift was recorded as the 1-RM. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Percentage change from Baseline was calculated by 100*[(post-dose value minus Baseline value)/ Baseline value]. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 20 | 18 | 21 | 21
Percentage change | 0.08 (2.787) | 16.78 (2.925) | 5.73 (3.921) | 11.07 (3.922)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 16.71, 90% CI 2-sided [9.86 to 23.56] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 5.35, 90% CI 2-sided [-4.09 to 14.78] — [estimate comment as in outcome 14, analysis 1]

16. Primary Outcome: Percentage Change From Baseline in Maximum Leg Press Strength Following 1 Repetition Maximum (1-RM) at Day 90
Description: as for outcome 15
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 19 | 18 | 18 | 20
Percentage change | 12.76 (4.061) | 17.93 (4.179) | 7.15 (2.759) | 14.17 (2.632)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 5.17, 90% CI 2-sided [-4.67 to 15.01] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 7.02, 90% CI 2-sided [0.46 to 13.58] — [estimate comment as in outcome 14, analysis 1]

17. Primary Outcome: Change From Baseline in Maximum Leg Press Strength Following 1 Repetition Maximum (1-RM) at Day 28
Description: Lower extremity strength was measured as 1-RM on a leg press device. Participants continued with a one set of 5 to 10 repetitions of lifting weights using 40 to 60% of estimated maximum, after warm up. Participants, then lifted progressively heavier weights in steps, with each step separated by an appropriate rest period, until participant could not complete the lift. The last successfully completed lift was recorded as the 1-RM. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 28
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 20 | 22 | 23
Kilograms | 4.2 (3.01) | 10.0 (3.08) | 3.0 (5.06) | 16.5 (4.90)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 5.9, 90% CI 2-sided [-1.4 to 13.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 13.5, 90% CI 2-sided [1.6 to 25.5] — [estimate comment as in outcome 14, analysis 1]

18. Primary Outcome: Change From Baseline in Maximum Leg Press Strength Following 1 Repetition Maximum (1-RM) at Day 56
Description: as for outcome 17
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 20 | 18 | 21 | 21
Kilograms | 0.6 (4.29) | 21.3 (4.50) | 8.3 (7.69) | 15.7 (7.69)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 20.7, 90% CI 2-sided [10.1 to 31.2] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 7.3, 90% CI 2-sided [-11.1 to 25.8] — [estimate comment as in outcome 14, analysis 1]

19. Primary Outcome: Change From Baseline in Maximum Leg Press Strength Following 1 Repetition Maximum (1-RM) at Day 90
Description: as for outcome 17
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 19 | 18 | 18 | 20
Kilograms | 12.3 (4.31) | 20.3 (4.45) | 14.2 (5.17) | 26.0 (4.91)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 8.0, 90% CI 2-sided [-2.5 to 18.4] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 11.8, 90% CI 2-sided [-0.5 to 24.0] — [estimate comment as in outcome 14, analysis 1]

20. Secondary Outcome: Change From Baseline in Appendicular Lean Mass as Assessed by Dual-energy X-ray Absorptiometry (DXA) at Day 28
Description: Participants were asked to lie on a padded platform while a mechanical arm passed over their body. Appendicular lean mass was calculated from the regional lean mass measurements of the arms and legs using DXA. Day 1 (Pre-dose) was considered as a Baseline. Analysis was performed using mixed model repeated measures. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 28
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 20 | 22
Kilograms | -0.240 (0.0974) | 0.642 (0.1023) | 0.055 (0.1920) | 0.346 (0.1831)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 0.882, 90% CI 2-sided [0.643 to 1.121] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and Baseline appendicular lean mass, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 0.291, 90% CI 2-sided [-0.156 to 0.738] — [estimate comment as in outcome 20, analysis 1]

21. Secondary Outcome: Change From Baseline in Appendicular Lean Mass as Assessed by Dual-energy X-ray Absorptiometry (DXA) at Day 56
Description: as for outcome 20
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 17 | 18
Kilograms | -0.134 (0.1410) | 0.848 (0.1540) | -0.464 (0.1887) | 0.663 (0.1829)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 0.982, 90% CI 2-sided [0.629 to 1.334] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 1.127, 90% CI 2-sided [0.682 to 1.571] — [estimate comment as in outcome 20, analysis 1]

22. Secondary Outcome: Change From Baseline in Appendicular Lean Mass as Assessed by Dual-energy X-ray Absorptiometry (DXA) at Day 90
Description: as for outcome 20
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 15 | 18
Kilograms | -0.434 (0.1657) | 0.946 (0.1818) | -0.225 (0.2306) | 0.899 (0.2117)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 1.380, 90% CI 2-sided [0.964 to 1.795] — [estimate comment as in outcome 20, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 1.124, 90% CI 2-sided [0.594 to 1.654] — [estimate comment as in outcome 20, analysis 1]

23. Secondary Outcome: Change From Baseline in Total Lean Mass as Assessed by Dual-energy X-ray Absorptiometry (DXA) at Day 28
Description: Participants were asked to lie on a padded platform while a mechanical arm passed over their body. Total lean mass was measured using DXA. Day 1 (Pre-dose) was considered as a Baseline. Analysis was performed using mixed model repeated measures. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 28
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 20 | 22
Kilograms | -0.017 (0.2004) | 1.150 (0.2106) | 0.075 (0.3004) | 0.998 (0.2869)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 1.167, 90% CI 2-sided [0.677 to 1.658] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and Baseline total lean mass, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 0.923, 90% CI 2-sided [0.222 to 1.623] — [estimate comment as in outcome 23, analysis 1]

24. Secondary Outcome: Change From Baseline in Total Lean Mass as Assessed by Dual-energy X-ray Absorptiometry (DXA) at Day 56
Description: as for outcome 23
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 17 | 18
Kilograms | -0.564 (0.2372) | 1.522 (0.2587) | -0.373 (0.3820) | 1.327 (0.3700)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 2.085, 90% CI 2-sided [1.493 to 2.678] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 1.700, 90% CI 2-sided [0.801 to 2.600] — [estimate comment as in outcome 23, analysis 1]

25. Secondary Outcome: Change From Baseline in Total Lean Mass as Assessed by Dual-energy X-ray Absorptiometry (DXA) at Day 90
Description: as for outcome 23
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 15 | 18
Kilograms | -0.531 (0.3349) | 1.577 (0.3666) | -0.424 (0.5056) | 1.689 (0.4666)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 2.108, 90% CI 2-sided [1.271 to 2.945] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 2.113, 90% CI 2-sided [0.949 to 3.277] — [estimate comment as in outcome 23, analysis 1]

26. Secondary Outcome: Change From Baseline in Total Short Physical Performance Battery (SPPB) Score at Day 28
Description: Participants were assessed for balance, time for chair rise and gait speed. These are the three components of SPPB. Each component was scored from 0 to 4. The total SPPB score was calculated by taking sum of scores of all 3 components, which ranged from 0 (worst performance) to 12 (best performance). Higher scores indicated better performance. Scores 10 to 12 indicated 'fit/normal' and scores <=7 indicated frail participant. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 28
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 20 | 22 | 23
Scores on a scale | 0.3 (0.25) | 0.4 (0.26) | 0.2 (0.19) | 0.3 (0.18)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 0.0, 90% CI 2-sided [-0.6 to 0.6] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and Baseline SPPB total score, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 0.0, 90% CI 2-sided [-0.4 to 0.5] — [estimate comment as in outcome 26, analysis 1]

27. Secondary Outcome: Change From Baseline in Total Short Physical Performance Battery (SPPB) Score at Day 56
Description: as for outcome 26
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 21 | 21
Scores on a scale | 0.4 (0.24) | 0.4 (0.25) | 0.1 (0.24) | 0.4 (0.24)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 0.0, 90% CI 2-sided [-0.6 to 0.6] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 0.3, 90% CI 2-sided [-0.2 to 0.9] — [estimate comment as in outcome 26, analysis 1]

28. Secondary Outcome: Change From Baseline in Total Short Physical Performance Battery (SPPB) Score at Day 90
Description: as for outcome 26
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 18 | 18 | 20
Scores on a scale | 0.3 (0.26) | 0.5 (0.28) | 0.4 (0.23) | 0.5 (0.22)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 0.2, 90% CI 2-sided [-0.4 to 0.9] — [estimate comment as in outcome 26, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 0.1, 90% CI 2-sided [-0.5 to 0.6] — [estimate comment as in outcome 26, analysis 1]

29. Secondary Outcome: Change From Baseline in 'Time for Chair Rise' as Assessed by SPPB at Day 28
Description: 'Time for chair rise' is one of the 3 components of SPPB, which was assessed by repeated chair stand test and calculated as time for five successful chair stands measured in seconds. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Analysis was performed using mixed model repeated measures. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 28
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 20 | 22 | 23
Seconds | -0.644 (0.6333) | -1.196 (0.6491) | -0.464 (0.3841) | -0.537 (0.3763)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.553, 90% CI 2-sided [-2.082 to 0.977] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and corresponding Baseline time for chair rise, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -0.073, 90% CI 2-sided [-0.977 to 0.832] — [estimate comment as in outcome 29, analysis 1]

30. Secondary Outcome: Change From Baseline in 'Time for Chair Rise' as Assessed by SPPB at Day 56
Description: as for outcome 29
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 21 | 21
Seconds | -1.207 (0.5912) | -2.023 (0.6124) | -0.323 (0.5294) | -0.160 (0.5282)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.816, 90% CI 2-sided [-2.252 to 0.619] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 0.163, 90% CI 2-sided [-1.096 to 1.422] — [estimate comment as in outcome 29, analysis 1]

31. Secondary Outcome: Change From Baseline in 'Time for Chair Rise' as Assessed by SPPB at Day 90
Description: as for outcome 29
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 18 | 18 | 20
Seconds | -1.070 (0.6956) | -2.030 (0.7362) | 1.144 (1.4013) | -0.793 (1.3401)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.960, 90% CI 2-sided [-2.668 to 0.748] — [estimate comment as in outcome 29, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -1.937, 90% CI 2-sided [-5.208 to 1.333] — [estimate comment as in outcome 29, analysis 1]

32. Secondary Outcome: Change From Baseline in 'Time for Fastest Walk for 4 Meter' as Assessed by SPPB at Day 28
Description: ''Time for fastest walk for 4 meter' was assessed by SPPB using 4 meter gait speed test. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Analysis was performed using mixed model repeated measures. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 28
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 20 | 22 | 23
Seconds | -0.236 (0.1132) | -0.277 (0.1161) | -0.167 (0.1133) | -0.110 (0.1108)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.040, 90% CI 2-sided [-0.314 to 0.233] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and corresponding Baseline Time for fastest walk for 4 meter, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 0.058, 90% CI 2-sided [-0.209 to 0.324] — [estimate comment as in outcome 32, analysis 1]

33. Secondary Outcome: Change From Baseline in 'Time for Fastest Walk for 4 Meter' as Assessed by SPPB at Day 56
Description: 'Time for fastest walk for 4 meter' was assessed by SPPB using 4 meter gait speed test. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Analysis was performed using mixed model repeated measures. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 21 | 21
Seconds | 0.010 (0.1487) | -0.276 (0.1560) | -0.093 (0.1437) | -0.284 (0.1438)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.287, 90% CI 2-sided [-0.650 to 0.077] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -0.191, 90% CI 2-sided [-0.534 to 0.152] — [estimate comment as in outcome 32, analysis 1]

34. Secondary Outcome: Change From Baseline in 'Time for Fastest Walk for 4 Meter' as Assessed by SPPB at Day 90
Description: as for outcome 33
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 18 | 18 | 20
Seconds | -0.043 (0.2194) | -0.055 (0.2361) | -0.130 (0.1331) | -0.360 (0.1275)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.012, 90% CI 2-sided [-0.555 to 0.532] — [estimate comment as in outcome 32, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -0.231, 90% CI 2-sided [-0.541 to 0.080] — [estimate comment as in outcome 32, analysis 1]

35. Secondary Outcome: Change From Baseline in Constant Work Rate (CWR) Duration From Endurance Shuttle Walking Test
Description: The endurance shuttle walk test is a CWR test requiring the participant to walk around a flat 10 meter track at a constant individualized pace. The test was externally paced, set to elicit a maximal exercise response (pace was based on a fixed percentage of prior incremental shuttle walk test performance, which determined a participant's peak exercise capacity). CWR duration is the time in seconds required by a participant to cover a flat 10 meter track during this test. Day 1 (Pre-dose) was considered as a Baseline. Analysis was performed using analysis of covariance (ANCOVA) model. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Seconds
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 19 | 16 | 18 | 20
Seconds | -6.5 (26.78) | 4.6 (29.25) | 105.1 (54.94) | -44.2 (51.97)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Difference in Least Square Means = 11.1, 90% CI 2-sided [-57.1 to 79.2] — Analysis was performed by ANCOVA model with Baseline CWR duration as the covariate adjusting for the treatment
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Difference in Least Square Means = -149.3, 90% CI 2-sided [-280.6 to -18.1] — Analysis was performed by ANCOVA model with Baseline CWR duration as the covariate adjusting for the treatment

36. Secondary Outcome: Change From Baseline in Peak Performance From Incremental Shuttle Walking Test
Description: An incremental shuttle walk test is an externally paced maximal exercise test which determined a participant's peak exercise capacity. The maximum duration of the test is 20 minutes. Peak performance was measured in meters, which was defined as the maximum distance covered by a participant until the participant can no longer continue walking during this test. Baseline was defined as the highest non-missing pre-dose assessment from Day -9 and Day 1. Analysis was performed using ANCOVA model. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Highest non-missing pre-dose assessment from Day-9 and Day 1), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 19 | 18 | 18 | 20
Meters | -10.5 (14.76) | -17.2 (15.16) | -7.5 (15.84) | -42.3 (15.02)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Difference in Least Square Means = -6.7, 90% CI 2-sided [-42.7 to 29.2] — Analysis was performed by ANCOVA model with Baseline peak performance as the covariate adjusting for the treatment
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Difference in Least Square Means = -34.8, 90% CI 2-sided [-72.0 to 2.4] — Analysis was performed by ANCOVA model with Baseline peak performance as the covariate adjusting for the treatment

37. Secondary Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) Score at Day 56
Description: The CAT is a short and simple participant-completed questionnaire which was developed for use in routine clinical practice to measure the health status of participants with COPD. The CAT is an 8-item questionnaire suitable for completion by all participants diagnosed with COPD. Participants rated their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment). A total CAT score was calculated by summing the non-missing scores of the eight items with a scoring range of 0-40. Higher scores indicated more severe disease impact. Day 1 (Pre-dose) was considered as a Baseline. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented.
Time Frame: Baseline (Day 1, Pre-dose), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 21 | 21
Scores on a Scale | -0.8 (0.92) | -1.2 (0.97) | -0.4 (1.14) | -1.0 (1.14)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.4, 90% CI 2-sided [-2.6 to 1.9] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and Baseline CAT score, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -0.7, 90% CI 2-sided [-3.4 to 2.1] — [estimate comment as in outcome 37, analysis 1]

38. Secondary Outcome: Change From Baseline in Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) Score at Day 90
Description: as for outcome 37
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 18 | 18 | 20
Scores on a Scale | -1.3 (0.79) | -2.2 (0.85) | -1.4 (0.94) | 0.8 (0.90)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -0.9, 90% CI 2-sided [-2.9 to 1.1] — [estimate comment as in outcome 37, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 2.2, 90% CI 2-sided [0.0 to 4.5] — [estimate comment as in outcome 37, analysis 1]

39. Secondary Outcome: Change From Baseline in Participant Reported Outcome (PRO)Active Individual Component: Difficulty Score at Day 56
Description: The daily PROactive instrument consisted of a PRO questionnaire and an activity monitor to measure participant experience of physical activity. It consisted of 9-item daily assessments covering 2 different domains (amount and difficulty). The 'amount' domain was covered by 2 questions combined with 2 activity monitor outputs. The 'difficulty' domain was covered by 5 questions. Individual domains were scored by simple adding items, gave raw score values 0 to 17 for 'amount' and 0 to 20 for 'difficulty'. The raw scores were then transformed to a 0 to 100 Rasch analysis based scale for each domain. Higher scores indicated worse experience with physical activity. Baseline was the average of the data collected from the 7-day period after dispensing of the device on Day -9. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented for averaged weekly difficulty score.
Time Frame: Baseline (Day -9), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 17 | 12 | 12 | 13
Scores on a Scale | 3.7 (1.59) | -1.1 (1.80) | 1.3 (2.16) | -0.8 (2.08)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -4.7, 90% CI 2-sided [-8.9 to -0.6] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and corresponding Baseline difficulty scores, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -2.1, 90% CI 2-sided [-7.2 to 3.1] — [estimate comment as in outcome 39, analysis 1]

40. Secondary Outcome: Change From Baseline in Participant Reported Outcome (PRO)Active Individual Component: Difficulty Score at Day 90
Description: as for outcome 39
Time Frame: Baseline (Day -9), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 15 | 17 | 13 | 11
Scores on a Scale | 2.0 (1.90) | -2.9 (1.84) | 2.8 (2.56) | -1.2 (2.65)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -4.9, 90% CI 2-sided [-9.5 to -0.4] — [estimate comment as in outcome 39, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -4.1, 90% CI 2-sided [-10.3 to 2.2] — [estimate comment as in outcome 39, analysis 1]

41. Secondary Outcome: Change From Baseline in Participant Reported Outcome (PRO)Active Individual Component: Amount Score at Day 56
Description: The daily PROactive instrument consisted of a PRO questionnaire and an activity monitor to measure participant experience of physical activity. It consisted of 9-item daily assessments covering 2 different domains (amount and difficulty). The 'amount' domain was covered by 2 questions combined with 2 activity monitor outputs. The 'difficulty' domain was covered by 5 questions. Individual domains were scored by simple adding items, gave raw score values 0 to 17 for 'amount' and 0 to 20 for 'difficulty'. The raw scores were then transformed to a 0 to 100 Rasch analysis based scale for each domain. Higher scores indicated worse experience with physical activity. Baseline was the average of the data collected from the 7-day period after dispensing of the device on Day -9. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented for averaged weekly amount score.
Time Frame: Baseline (Day -9), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 17 | 12 | 12 | 13
Scores on a Scale | 3.3 (1.09) | 0.2 (1.24) | 2.5 (1.83) | 2.3 (1.77)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -3.1, 90% CI 2-sided [-5.9 to -0.3] — Analysis was performed by mixed model repeated measures including the covariates: treatment, Day, treatment*Day and corresponding Baseline amount scores, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -0.2, 90% CI 2-sided [-4.6 to 4.2] — [estimate comment as in outcome 41, analysis 1]

42. Secondary Outcome: Change From Baseline in Participant Reported Outcome (PRO)Active Individual Component: Amount Score at Day 90
Description: as for outcome 41
Time Frame: Baseline (Day -9), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 15 | 17 | 13 | 11
Scores on a Scale | -0.2 (2.05) | 3.8 (1.98) | -0.8 (2.33) | 2.7 (2.47)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = 4.0, 90% CI 2-sided [-0.8 to 8.8] — [estimate comment as in outcome 41, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = 3.5, 90% CI 2-sided [-2.3 to 9.4] — [estimate comment as in outcome 41, analysis 1]

43. Secondary Outcome: Change From Baseline in Participant Reported Outcome (PRO)Active Total Score at Day 56
Description: The daily PROactive instrument consisted of a PRO questionnaire and an activity monitor to measure participant experience of physical activity. It consisted of 9-item daily assessments covering 2 different domains(amount and difficulty). The'amount'domain was covered by 2 questions combined with 2 activity monitor outputs. The 'difficulty'domain was covered by 5 questions. Individual domains were scored by simple adding items, gave raw score values 0 to 17 for'amount'and 0 to 20 for'difficulty. The raw scores were then transformed to a 0 to 100 Rasch scale for each domain. The 'total score' was obtained by calculating the average between two domains. Total score has the range from 0 to 100. Higher scores indicated worse experience with physical activity. Baseline was the average of the data collected from the 7-day period after dispensing of the device on Day -9. Change from Baseline was calculated as post-dose visit value minus the Baseline value. Adjusted means and SE are presented
Time Frame: Baseline (Day -9), Day 56
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 17 | 12 | 12 | 13
Scores on a Scale | 3.7 (0.89) | -0.5 (1.03) | 2.1 (1.09) | 0.5 (1.05)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -4.2, 90% CI 2-sided [-6.5 to -1.9] — Analysis was performed by mixed model repeated measures including the covariates; treatment, Day, treatment*Day and corresponding Baseline total scores, with Day as the repeated factor
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -1.5, 90% CI 2-sided [-4.1 to 1.1] — [estimate comment as in outcome 43, analysis 1]

44. Secondary Outcome: Change From Baseline in Participant Reported Outcome (PRO)Active Total Score at Day 90
Description: as for outcome 43
Time Frame: Baseline (Day -9), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 15 | 17 | 13 | 11
Scores on a Scale | 1.3 (1.20) | 0.3 (1.14) | 1.2 (1.57) | 0.5 (1.66)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Mean Difference (Net) = -1.0, 90% CI 2-sided [-3.8 to 1.8] — [estimate comment as in outcome 43, analysis 1]
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Mean Difference (Net) = -0.7, 90% CI 2-sided [-4.6 to 3.2] — [estimate comment as in outcome 43, analysis 1]

45. Secondary Outcome: Change From Baseline in Steps Per Day (Physical Activity Measure) as Assessed Via an Accelerometer
Description: Steps per day was assessed using an accelerometer, a clinically validated physical activity monitor which was used to measure the levels of physical activity. Participants wore an accelerometer for 7 days during individual timepoint. Values at Baseline, Day 56 and Day 90 were the average values collected from an accelerometer for 7 days after the Day -9, Day 56 and Day 90. Baseline was the average of the data collected from the 7-day period after dispensing of the device on Day -9. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day -9), Days 56 and 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Steps per day
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 17 | 17 | 14 | 17
Steps per day
  Day 56,n=17,14,14,17: number analyzed (Participants) | 17 | 14 | 14 | 17
  Day 56,n=17,14,14,17 | 285.19 (1289.604) | 389.58 (1322.701) | 120.41 (1282.092) | -17.40 (1334.539)
  Day 90,n=17,17,14,14: number analyzed (Participants) | 17 | 17 | 14 | 14
  Day 90,n=17,17,14,14 | -246.45 (756.414) | 786.21 (1439.988) | -527.07 (1077.747) | 611.36 (1499.559)

46. Secondary Outcome: Change From Baseline in Vector Magnitude Unit Per Wear Time (Physical Activity Measure) as Assessed Via an Accelerometer
Description: Vector magnitude unit per wear time was assessed using an accelerometer, a clinically validated physical activity monitor which was used to measure the levels of physical activity. Participants wore an accelerometer for 7 days during individual timepoint. Values at Baseline, Day 56 and Day 90 were the average values collected from accelerometer for 7 days after the Day -9, Day 56 and Day 90. Data from an accelerator was uploaded to a central site. Baseline was the average of the data collected from the 7-day period after dispensing of the device on Day -9. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day -9), Days 56 and 90
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Vector magnitude units per minute
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 17 | 17 | 14 | 17
Vector magnitude units per minute
  Day 56,n=17,14,14,17: number analyzed (Participants) | 17 | 14 | 14 | 17
  Day 56,n=17,14,14,17 | 9.19 (82.596) | -4.83 (66.400) | 56.42 (86.284) | 71.98 (175.403)
  Day 90,n=17,17,14,14: number analyzed (Participants) | 17 | 17 | 14 | 14
  Day 90,n=17,17,14,14 | -6.60 (65.648) | 0.40 (64.670) | -3.73 (74.849) | 42.36 (184.191)

47. Secondary Outcome: Number of Participants With Participant Global Impression of Change (PGIC) Score Over Time
Description: Participant-reported response to treatment was assessed using the PGIC measure, a single item completed by participant to assess the participant's impression of change in their disease severity since the beginning of the study. Responses to the PGIC question were on a 7 point Likert scale: Much Better, Better, Slightly Better, No Change, Slightly Worse, Worse, and Much Worse. Number of participants with PGIC score is presented by treatment group, visit and by 7 response categories.
Time Frame: Days 14, 28, 56 and 90
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 20 | 23 | 23
Participants
  Day 14, much worse,n=21,20,23,23 | 0 | 0 | 0 | 0
  Day 14, worse,n=21,20,23,23 | 0 | 0 | 0 | 1
  Day 14, slightly worse,n=21,20,23,23 | 0 | 1 | 0 | 0
  Day 14, no change,n=21,20,23,23 | 6 | 5 | 9 | 9
  Day 14, slightly better,n=21,20,23,23 | 7 | 7 | 4 | 4
  Day 14, better,n=21,20,23,23 | 7 | 5 | 8 | 7
  Day 14, much better,n=21,20,23,23 | 1 | 2 | 2 | 2
  Day 28, much worse,n=21,20,21,22: number analyzed (Participants) | 21 | 20 | 21 | 22
  Day 28, much worse,n=21,20,21,22 | 0 | 0 | 0 | 0
  Day 28, worse,n=21,20,21,22: number analyzed (Participants) | 21 | 20 | 21 | 22
  Day 28, worse,n=21,20,21,22 | 0 | 0 | 0 | 0
  Day 28, slightly worse,n=21,20,21,22: number analyzed (Participants) | 21 | 20 | 21 | 22
  Day 28, slightly worse,n=21,20,21,22 | 1 | 2 | 0 | 0
  Day 28, no change,n=21,20,21,22: number analyzed (Participants) | 21 | 20 | 21 | 22
  Day 28, no change,n=21,20,21,22 | 3 | 6 | 4 | 6
  Day 28, slightly better,n=21,20,21,22: number analyzed (Participants) | 21 | 20 | 21 | 22
  Day 28, slightly better,n=21,20,21,22 | 9 | 6 | 10 | 7
  Day 28, better,n=21,20,21,22: number analyzed (Participants) | 21 | 20 | 21 | 22
  Day 28, better,n=21,20,21,22 | 5 | 6 | 5 | 7
  Day 28, much better,n=21,20,21,22: number analyzed (Participants) | 21 | 20 | 21 | 22
  Day 28, much better,n=21,20,21,22 | 3 | 0 | 2 | 2
  Day 56, much worse,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  Day 56, much worse,n=21,19,21,21 | 0 | 0 | 0 | 0
  Day 56, worse,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  Day 56, worse,n=21,19,21,21 | 0 | 0 | 0 | 0
  Day 56, slightly worse,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  Day 56, slightly worse,n=21,19,21,21 | 1 | 3 | 1 | 4
  Day 56, no change,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  Day 56, no change,n=21,19,21,21 | 2 | 5 | 4 | 5
  Day 56, slightly better,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  Day 56, slightly better,n=21,19,21,21 | 6 | 4 | 7 | 5
  Day 56, better,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  Day 56, better,n=21,19,21,21 | 10 | 6 | 8 | 5
  Day 56, much better,n=21,19,21,21: number analyzed (Participants) | 21 | 19 | 21 | 21
  Day 56, much better,n=21,19,21,21 | 2 | 1 | 1 | 2
  Day 90, much worse,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, much worse,n=21,18,18,20 | 0 | 0 | 0 | 0
  Day 90, worse,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, worse,n=21,18,18,20 | 0 | 1 | 0 | 0
  Day 90, slightly worse,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, slightly worse,n=21,18,18,20 | 1 | 0 | 0 | 0
  Day 90, no change,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, no change,n=21,18,18,20 | 9 | 8 | 5 | 6
  Day 90, slightly better,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, slightly better,n=21,18,18,20 | 7 | 3 | 9 | 9
  Day 90, better,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, better,n=21,18,18,20 | 3 | 4 | 4 | 4
  Day 90, much better,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, much better,n=21,18,18,20 | 1 | 2 | 0 | 1

48. Secondary Outcome: Number of Participants With Participant Global Rating of Severity (PGRS) Score Over Time
Description: PGRS is a single global question and was asked to participants to rate their COPD severity on a four point scale ranging from 1 to 4 (1=mild, 2=moderate, 3=severe, 4=very severe). Number of participants with PGRS score ranging from mild to very severe are presented over time.
Time Frame: Days 1 and 90
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 20 | 23 | 23
Participants
  Day 1, mild,n=21,20,23,23 | 2 | 0 | 0 | 2
  Day 1, moderate,n=21,20,23,23 | 9 | 13 | 11 | 12
  Day 1, severe,n=21,20,23,23 | 8 | 7 | 12 | 8
  Day 1, very severe,n=21,20,23,23 | 2 | 0 | 0 | 1
  Day 90, mild,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, mild,n=21,18,18,20 | 4 | 4 | 1 | 5
  Day 90, moderate,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, moderate,n=21,18,18,20 | 9 | 7 | 9 | 2
  Day 90, severe,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, severe,n=21,18,18,20 | 6 | 6 | 8 | 12
  Day 90, very severe,n=21,18,18,20: number analyzed (Participants) | 21 | 18 | 18 | 20
  Day 90, very severe,n=21,18,18,20 | 2 | 1 | 0 | 1

49. Secondary Outcome: Change From Baseline in St. George Respiratory Questionnaire (SGRQ) for COPD (SGRQ-c) Total Score
Description: SGRQ-c is the COPD specific version of SGRQ. It consisted of 40 items in total, corresponding to 3 individual domains (components): symptoms, activity and impact, with different components carrying a different weighting. Component scores were calculated by summing the weights from all positive items in that component, dividing by the sum of maximum possible weights for all items in that component, and multiplying this number by 100. Total score was calculated by summing the weight to all the positive responses in each component. Total score has the range from 0 to 100. Higher scores indicated more severe disease impact. Day 1 (Pre-dose) was considered as a Baseline. Analysis was performed using ANCOVA model. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 18 | 20
Scores on a scale | -3.9 (1.71) | -0.9 (1.90) | -1.7 (1.87) | 0.4 (1.77)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Difference in Least Square Means = 3.0, 90% CI 2-sided [-1.4 to 7.4] — Analysis was performed by ANCOVA model with Baseline total score as the covariate adjusting for the treatment
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Difference in Least Square Means = 2.1, 90% CI 2-sided [-2.3 to 6.5] — Analysis was performed by ANCOVA model with Baseline total score as the covariate adjusting for the treatment

50. Secondary Outcome: Change From Baseline in SGRQ-c Symptoms Score
Description: SGRQ-c is the COPD specific version of SGRQ. It consisted of 40 items in total, corresponding to 3 individual domains (components): symptoms, activity and impact, with different components carrying a different weighting. Component scores were calculated by summing the weights from all positive items in that component, dividing by the sum of maximum possible weights for all items in that component, and multiplying this number by 100. Symptoms component consisted of questions 1 to 7 in Part 1. Symptoms score has the range from 0 to 100. Higher scores indicated more severe disease impact. Day 1 (Pre-dose) was considered as a Baseline. Analysis was performed using ANCOVA model. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 18 | 20
Scores on a scale | -4.0 (2.95) | -1.4 (3.29) | -3.5 (3.38) | -4.0 (3.20)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Difference in Least Square Means = 2.6, 90% CI 2-sided [-5.0 to 10.1] — Analysis was performed by ANCOVA model with Baseline symptoms score as the covariate adjusting for the treatment
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Difference in Least Square Means = -0.5, 90% CI 2-sided [-8.4 to 7.5] — Analysis was performed by ANCOVA model with Baseline symptoms score as the covariate adjusting for the treatment

51. Secondary Outcome: Change From Baseline in SGRQ-c Activity Score
Description: SGRQ-c is the COPD specific version of SGRQ. It consisted of 40 items in total, corresponding to 3 individual domains (components): symptoms, activity and impact, with different components carrying a different weighting. Component scores were calculated by summing the weights from all positive items in that component, dividing by the sum of maximum possible weights for all items in that component, and multiplying this number by 100. Activity component consisted of questions 9 and 12 in Part 2 of the questionnaire. Activity score has the range from 0 to 100. Higher scores indicated more severe disease impact. Day 1 (Pre-dose) was considered as a Baseline. Analysis was performed using ANCOVA model. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 18 | 20
Scores on a scale | -5.4 (2.00) | -3.4 (2.23) | 1.2 (2.57) | 1.6 (2.44)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Difference in Least Square Means = 2.0, 90% CI 2-sided [-3.2 to 7.1] — Analysis was performed by ANCOVA model with Baseline activity score as the covariate adjusting for the treatment
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Difference in Least Square Means = 0.5, 90% CI 2-sided [-5.6 to 6.5] — Analysis was performed by ANCOVA model with Baseline activity score as the covariate adjusting for the treatment

52. Secondary Outcome: Change From Baseline in SGRQ-c Impact Score
Description: SGRQ-c is the COPD specific version of SGRQ. It consisted of 40 items in total, corresponding to 3 individual domains (components): symptoms, activity and impact, with different components carrying a different weighting. Component scores were calculated by summing the weights from all positive items in that component, dividing by the sum of maximum possible weights for all items in that component, and multiplying this number by 100. Impact component consisted of questions 8, 10, 11, 13, 14 in Part 2 of the questionnaire. Impact score has the range from 0 to 100. Higher scores indicated more severe disease impact. Day 1 (Pre-dose) was considered as a Baseline. Analysis was performed using ANCOVA model. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Day 90
Population: Analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 17 | 18 | 20
Scores on a scale | -2.8 (2.03) | 0.6 (2.25) | -2.7 (1.76) | 0.8 (1.67)
Statistical Analysis 1: Comparison: Placebo- Female Participants vs GSK2881078 1.0 mg- Female Participants; Test type: Other; Difference in Least Square Means = 3.4, 90% CI 2-sided [-1.7 to 8.6] — Analysis was performed by ANCOVA model with Baseline impact score as the covariate adjusting for the treatment
Statistical Analysis 2: Comparison: Placebo- Male Participants vs GSK2881078 2.0 mg- Male Participants; Test type: Other; Difference in Least Square Means = 3.5, 90% CI 2-sided [-0.7 to 7.7] — Analysis was performed by ANCOVA model with Baseline impact score as the covariate adjusting for the treatment

53. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FEV1 measurements were collected using a spirometer. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 56 and 90
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 21 | 21
Liters
  Day 56,n=21,19,21,21 | -0.000 (0.0918) | -0.028 (0.0747) | 0.012 (0.1342) | -0.016 (0.2377)
  Day 90,n=20,18,18,20: number analyzed (Participants) | 20 | 18 | 18 | 20
  Day 90,n=20,18,18,20 | 0.002 (0.0970) | -0.024 (0.0833) | 0.050 (0.1130) | 0.007 (0.2208)

54. Secondary Outcome: Change From Baseline in Sniff Nasal Inspiratory Pressure (SnIP)
Description: A bung size-specific to the participant was placed in the nostril deemed to be most patent by the investigator. The participant was asked to make a maximum voluntary sniff effort via a peak flow meter and the greatest effort from 10 repeat measurements were recorded. SnIP was measured in centimeter of water (cm H2O). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Days 56 and 90
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: centimeter of water
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 19 | 21 | 21
centimeter of water
  Day 56,n=21,19,21,21 | -6.0 (11.20) | 3.4 (14.14) | 0.7 (17.82) | -0.8 (15.51)
  Day 90,n=20,18,18,20: number analyzed (Participants) | 20 | 18 | 18 | 20
  Day 90,n=20,18,18,20 | -0.7 (8.55) | -0.4 (11.34) | -1.2 (15.21) | 2.5 (21.39)

55. Secondary Outcome: Clearance (CL) of GSK2881078 Following Oral Dose in Participants
Description: Blood samples were collected at designated timepoints. Pharmacokinetics (PK) parameters of GSK2881078 were calculated using non-compartmental methods.
Time Frame: Day 14 (Pre-dose), Day 28 (Pre-dose and at 1 to 4 hours Post-dose), Day 56 (at 5 to 8 hours Post-dose), Day 90 (Pre-dose)
Population: Pharmacokinetic Population comprised of participants in the 'All Participants (all randomized participants who received at least one dose of study medication)'' Population for whom a PK sample was obtained and analyzed for GSK2881078.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | GSK2881078 1.0 mg- Female Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 24
Liters per hour | 0.393 (59.5) | 0.476 (44.0)

56. Secondary Outcome: Volume of Distribution at Steady State (Vss) of GSK2881078 Following Oral Dose in Participants
Description: Blood samples were collected at designated timepoints. PK parameters of GSK2881078 were calculated using non-compartmental methods.
Time Frame: as for outcome 55
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | GSK2881078 1.0 mg- Female Participants | GSK2881078 2.0 mg- Male Participants
Number analyzed (Participants) | 21 | 24
Liters | 39.4 (16.3) | 48.3 (29.8)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until up to Day 132
Description: SAEs and non-serious AEs were reported for the Safety Population which comprised of all randomized participants who received at least one dose of study medication. This population was based on the treatment the participant received.
Arm/Group | Placebo- Female Participants | GSK2881078 1.0 mg- Female Participants | Placebo- Male Participants | GSK2881078 2.0 mg- Male Participants
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/24 | 2/24 | 0/25
Other Adverse Events (participants affected / at risk) | 15/23 | 18/24 | 13/24 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo- Female Participants (N=23) | GSK2881078 1.0 mg- Female Participants (N=24) | Placebo- Male Participants (N=24) | GSK2881078 2.0 mg- Male Participants (N=25)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo- Female Participants (N=23) | GSK2881078 1.0 mg- Female Participants (N=24) | Placebo- Male Participants (N=24) | GSK2881078 2.0 mg- Male Participants (N=25)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (8) | 2 (2) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 2 (3) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT03359473/SAP_000.pdf
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03359473/Prot_001.pdf